CLINICAL TRIAL: NCT02841449
Title: The Effect of Hydration Status on Glycemic Control and Appetite Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: University of Bristol (Other); Loughborough University (Other); European Hydration Institute (Other); Economic and Social Research Council, United Kingdom (Other); Lund University (Other)
Responsible Party: Principal Investigator, Harriet Carroll, PhD Student, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16/SW/0057
Record Dates: First submitted 2016-07-07; First posted 2016-07-22 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: Hydration; Glycemic control; Appetite; Endocrinology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypohydrated (Experimental): After being dehydrated in the heat tent, participants in this trial arm will be given 3 mL/kg lean body mass to consume over the rest of the day (e.g. a 75 kg participant with a body composition of 85 % fat free mass would consume 191 mL water [63.75 kg * 3 mL])
  Interventions: Behavioral: Hypohydrated
- Rehydrated (Experimental): After being dehydrated in the heat tent, participants in this trial arm will be given 40 mL/kg lean body mass plus 150 % of their water losses (from the heat tent procedure) over the rest of the day (e.g. a 75 kg participant with a body composition of 85 % fat free mass and lost 1 % of their body mass in the heat tent (0.75 kg) would consume 2550 mL [63.75 kg * 40 mL] + 1125 mL [750 g * 1.5], totalling 3675 mL).
  Interventions: Behavioral: Rehydrated

INTERVENTIONS:
Behavioral: Hypohydrated — Participants remain hypohydrated after the heat tent procedure
  Arms: Hypohydrated
Behavioral: Rehydrated — Participants rehydrate after the heat tent procedure
  Arms: Rehydrated

SUMMARY:
The aim of this study is to investigate whether hydration status affects blood sugar control and appetite regulation. In order to do this, participants will undergo a monitoring phase whereby their weight, diet and physical activity are monitored, followed by a dehydration protocol involving fluid restriction and sitting in a heat tent. In one arm of the trial, participants will remain dehydrated for the remainder of the day (i.e. after the heat tent) by having their fluid intake restricted, and in the other arm of the trial, participants will be rehydrated by consuming the necessary amount of plain water. All participants will undergo both arms of the trial, the order of which will be chosen randomly.

Several measures will be taken throughout the trial. Before participants go into the heat tent, they will provide a urine sample (for baseline hydration status as indicated by urine osmolality), a blood sample (for glucose, insulin, arginine vasopressin,/copeptin, ghrelin and serum osmolality and plasma volume), and have a peripheral quantitative computer tomography scan of their thigh to indicate muscle size. On the day proceeding the heat tent, participants will have these measures repeated, along with metabolic rate before consuming a 75 g glucose drink, followed by 15 minutely blood samples and hourly metabolic rate measures for 120 minutes (i.e. an oral glucose tolerance test; OGTT). Following this, participants will be presented with a large bowl of pasta and sauce and will be instructed to eat until satisfied (maximum 30 min). Blood samples will be taken every 10 minutes for 60 minutes following the meal.

Participants also have the option to opt-in to have a muscle biopsy taken. This will be taken before and ~120 minutes after the glucose drink.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether hydration status affects blood sugar control and appetite regulation. This will be a randomised crossover trial with two trial arms separated by 5-35 days. Each trial arm consists of five days in total, with the only difference between the trial arms being the amount of fluid consumed after the heat tent on day 4 (as described below).

Days 1-3 of each trial arm are the monitoring phase. Participants will be given a chest mounted activity monitor (ActiHeart TM), some body mass scales, a food diary with food weighing scales and three urine sample pots. Participants will be required to provide a urine sample upon waking, and note their weight before eating. The activity monitor will need to be worn from midnight on day 1 in order to gauge three full 24-h periods of activity. The food diary will also start at this point; participants will be required to weigh and record all their food and beverages (including recording the leftovers). On day 3 of the monitoring phase, participants will be required to continue their normal daily routine, however they will be provided with a set amount of water to consume (40 mL/kg lean body mass) in order to standardize baseline hydration status. No food or fluid will be allowed to be consumed after 2200 h on day 3.

On day 4, participants will take the same measures (weight and urine sample) and will arrive at the university in a fasted state (i.e. no food or fluid). A blood sample will be drawn from an antecubital vein followed by a peripheral quantitative computer tomography (pQCT) scan of the thigh. After the blood sample and scan, participants may eat food from a list of low water-content foods only for the rest of the day. At approximately midday (flexible depending on the participants' availability, but matched on both trial arms), participants will be weighed again, and placed in a heat tent (40-50 degrees Celsius) until they lose 1 % of their pre-heat tent weight or for a maximum of one hour (whichever comes first). On the second trial arm, participants will be matched by percentage of body mass loss, even if this requires spending more or less time in the heat tent, but still no more than one hour.

After the heat tent, participants will receive a salty meal in order to facilitate fluid absorption/retention. This will be matched in both trial arms in order to reduce confounding. In the dehydration trial arm, participants will be provided with 3 mL/kg lean body mass of plain water to consume for the rest of the day. In the rehydration trial arm, participants will be given 40 mL/kg lean body mass plus 150 % of their body mass losses from the heat tent. This will be metered out throughout the day to maximise rehydration. Thus the amount of water consumed on day 4 after the heat tent is the only discernible difference between the trial arms, with everything else matched. In both trial arms only plain water (i.e. no caffeine or alcohol) will be allowed to be consumed, and only foods from the dry food list can be eaten. This will be matched on the subsequent trial arm. No food or fluid after 2200 h on day 4.

On the fifth day of each trial arm, participants will be required to attend the laboratory at approximately 0730 h (± 1 h). A urine sample will be collected, along with body mass. Another pQCT scan of the thigh will be taken and participants' metabolic rate will be measured using the Douglas bag method. As part of the trial, participants are able to opt-in for a muscle biopsy. If they have opted-in, a muscle biopsy will be taken after the pQCT scan. This will involve a local anesthetic (Lidocaine), making a small incision using a scalpel, then obtaining a muscle sample using the Bergstrom technique. Participants will then be fitted with a cannula, and their hand will be placed in a 60 degree Celsius hotbox for five minutes, after which a baseline blood sample will be drawn. Participants will be given a 75 g glucose drink to consume within five minutes. Whilst remaining rested, a researcher will draw a 10 mL blood sample every 15 minutes for 120 minutes, with approximately 10 mL saline infused after each blood sample drawn. Metabolic rate will be measured at 0 (pre-OGTT), 60 and 120 minutes. For the participants who opted-in for the muscle biopsy, another one will be taken after 120 minutes.

Participants will then be presented with some computer based appetite assessing psychological inventories to assess subconscious food preferences. These tests are pilot data for future research. Following this, participants will be presented with a pasta meal, with the instruction to eat until satisfied for a maximum of 30 minutes. After 30 minutes, a blood sample will be drawn, followed by 10 minutely samples for 60 minutes. Visual analogue scales for subjective appetite ratings will be taken pre-meal, immediately, post-meal, then at 30 and 60 minutes post-meal. The cannula will then be removed.

The sample size required for this trial is 16 participants, calculated using pilot data which assessed blood glucose control after being dehydrated and rehydrated. Based on that pilot study, hydration status resulted in a marked difference in the rate of return to fasted glycaemia. This primary conclusion was supported by a magnitude of effect 45 minutes post-oral glucose tolerance test (D = 1.1 mmol/l). The standard deviation at this time point in the control (normal hydration) group was also 1.1 mmol/l, resulting in an effect size (d) of ≈1. To provide a 95 % power (beta level) to detect this effect at an alpha level (p) of less than or equal to 0.05 using a 2--tailed paired t--test will require ~16 participants.

If any participant does not complete the study (i.e. they have missing data), their data will not be included in the analysis. In other words, the analysis plan will be per protocol (completers only). The statistical techniques used will be linear modelling with post-hoc t-tests corrected for multiple comparisons where relevant. However, until the final dataset has been obtained, the statistical tests may be subject to change (e.g. if data are non-parametric).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Aged 18-60 years
* Able and willing to give informed consent

Exclusion Criteria:

* Any known metabolic or glucose disorder
* Taking necessary medication (other than contraceptives) or supplements that are known to affect glycaemic control (e.g. chromium, PUFAs)
* Current alcohol or drug dependency
* Aged < 18 years, or > 60 years; pregnant or breastfeeding
* Any other factors which are deemed to have the potential to cause harm to the participant and/or could introduce bias into the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet A Carroll, MRes, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared
Supporting Information: Study Protocol, CSR
Time Frame: Available (no time restrictions)
Access Criteria: Open access; doi URL below for hydration-glycaemia data, related report: https://doi.org/10.1152/japplphysiol.00771.2018; data for hydration-appetite: https://doi.org/10.15125/BATH-00719 and related report: https://doi.org/10.1016/j.physbeh.2019.112725
URL: https://doi.org/10.15125/BATH-00547

REFERENCES:
- [Background] Taveau C, Chollet C, Waeckel L, Desposito D, Bichet DG, Arthus MF, Magnan C, Philippe E, Paradis V, Foufelle F, Hainault I, Enhorning S, Velho G, Roussel R, Bankir L, Melander O, Bouby N. Vasopressin and hydration play a major role in the development of glucose intolerance and hepatic steatosis in obese rats. Diabetologia. 2015 May;58(5):1081-90. doi: 10.1007/s00125-015-3496-9. Epub 2015 Jan 27. PMID 25622862
- [Background] Roussel R, Fezeu L, Bouby N, Balkau B, Lantieri O, Alhenc-Gelas F, Marre M, Bankir L; D.E.S.I.R. Study Group. Low water intake and risk for new-onset hyperglycemia. Diabetes Care. 2011 Dec;34(12):2551-4. doi: 10.2337/dc11-0652. Epub 2011 Oct 12. PMID 21994426
- [Background] Keller U, Szinnai G, Bilz S, Berneis K. Effects of changes in hydration on protein, glucose and lipid metabolism in man: impact on health. Eur J Clin Nutr. 2003 Dec;57 Suppl 2:S69-74. doi: 10.1038/sj.ejcn.1601904. PMID 14681716
- [Background] Zerbe RL, Vinicor F, Robertson GL. Plasma vasopressin in uncontrolled diabetes mellitus. Diabetes. 1979 May;28(5):503-8. doi: 10.2337/diab.28.5.503. PMID 108167

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: n = 17 recruited; n = 1 withdrew prior to starting the study due to surgery (unrelated to study)
Groups:
- Hypohydrated First, Then Rehydrated: After being dehydrated in the heat tent, participants in this trial arm will be given 3 mL/kg body mass to consume over the rest of the day (e.g. a 75 kg participantwould consume 225 mL water. After a 3-35 day washout, they will repeat the protocol but after the heat tent be given 40 mL/kg body mass + 150 % body mass losses from the heat tent in water.
  Hypohydrated: Participants remain hypohydrated after the heat tent procedure
- Rehydrated First, Then Hypohydrated: After being dehydrated in the heat tent, participants in this trial arm will be given 40 mL/kg body mass plus 150 % of their water losses (from the heat tent procedure) over the rest of the day (e.g. a 75 kg participant and lost 1 % of their body mass in the heat tent (0.75 kg) would consume 3000 mL + 1125 mL [750 g * 1.5], totalling 4125 mL). Following a 3-35 d washout, participants would then repeat the protocol but after the heat tent be given 3 mL/kg body mass of water to consume over the rest of the day.
  Rehydrated: Participants rehydrate after the heat tent procedure
Period: Overall Study
Arm/Group | Hypohydrated First, Then Rehydrated | Rehydrated First, Then Hypohydrated
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: crossover study; all participants did both arms of the trial
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypohydrated First, Then Rehydrated | Rehydrated First, Then Hypohydrated | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants] — Population: crossover study so participants all did both trial arms
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 7 | 9 | 16
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (8) | 31 (10) | 30 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Response
Description: Primary analysis is time trends (i.e. ANOVA effects), supported by indices of the glycemic response (e.g. iAUC, time to peak). Blood was taken pre-muscle biopsy (if participants opted in for a muscle biopsy), before consuming the glucose drink (after the biopsy, where applicable), then at 15 minutely samples for 120 minutes. After the meal test, blood was drawn at 10 minutely intervals for 60 minutes, starting 30 minutes after commencement of eating.
Time Frame: Measured on day 5 on both trial arms, using the blood sample drawn before the glucose beverage is consumed and the blood samples drawn for the subsequent 120 minutes
Measure: Mean (Standard Deviation); unit: mmol*120 min*l-1
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
mmol*120 min*l-1 | 303 (121) | 306 (113)
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.886, t-test, 2 sided; paired sample
Statistical Analysis 2: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.430, ANOVA — The above is the trial*time interaction. trial, p = 0.627; time, p < 0.001; repeated measures

2. Secondary Outcome: Insulinemic Response
Description: Primary analysis is time trends (i.e. ANOVA effects), supported by indices of the insulinemic response (e.g. iAUC, time to peak). Bloods drawn at pre-biopsy, pre-OGTT, 15, 30, 45, 60, 90, 120 min and 0, 30, 60 minutes after the ad libitum meal test.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol*120 min*l-1
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
pmol*120 min*l-1 | 20860 (8311) | 21937 (8340)
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.369, t-test, 2 sided; paired samples
Statistical Analysis 2: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.859, ANOVA — The above is the trial*time interaction. trial p = 0.200; time p < 0.001; repeated measures

3. Secondary Outcome: Arginine Vasopressin and Copeptin Response
Description: Primary analysis is time trends (i.e. ANOVA effects), supported by indices of the response trends (e.g. iAUC, time to peak). Bloods drawn pre-biopsy, pre-OGTT, and then 15 minutely for 120 minutes, and then 10 minutely after the ad libitum meal test.
Time Frame: Measured on day 5 on both trial arms, using the blood sample drawn before the glucose beverage is consumed and the blood samples drawn for the subsequent 120 minutes (please note: may measure copeptin as a marker of arginine vasopressin)
Measure: Mean (Standard Deviation); unit: pmol*120 min*l-1
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
pmol*120 min*l-1 | 2704 (2398) | 961 (1488)
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p < 0.001, t-test, 2 sided; paired samples
Statistical Analysis 2: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.261, ANOVA — The above is the trial*time interaction. trial p = 0.002; time p = 0.282; repeated measures

4. Secondary Outcome: Ghrelin Response
Description: Primary analysis is time trends (i.e. ANOVA effects), supported by indices of the response trend (e.g. iAUC, time to peak). Due to funding limitations, we only took one 60 minute postprandial measure of ghrelin.
Time Frame: Measured on day 5 on both trial arms, using the blood sample drawn before the participant starts eating the buffet and the subsequent post-buffet blood samples
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
pg/mL | 180 (65) | 188 (71)
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.736, t-test, 2 sided; paired samples

5. Secondary Outcome: Energy Intake
Description: Differences in energy intake between the hypohydrated and rehydrated groups (two-tailed t-test)
Time Frame: Measured on day 5 on both trial arms from the pasta test meal
Measure: Mean (Standard Deviation); unit: kJ
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
kJ | 1953 (742) | 2027 (926)
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.542, t-test, 2 sided; paired samples

6. Secondary Outcome: Metabolic Rate
Description: Comparing respiratory quotient and metabolic rate
Time Frame: Using the metabolic rate data collected on day 5 on both trial arms
Measure: Mean (Standard Deviation); unit: kJ*kg-1*day-1
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
kJ*kg-1*day-1 | 96.32 (11.94) | 95.11 (13.09)
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.400, t-test, 2 sided; paired samples

7. Secondary Outcome: Subjective Appetite Ratings
Description: Comparing appetite response. Scales were visual analogue scales of hunger, fullness, how much you feel you can eat, thirst, and desire for sweet, salty, savoury and fatty foods. Scales were 0-100 mm vertical lines which participants marked where 0 = not at all/no desire and 100 = extremely/very high desire)
Time Frame: Collected on day 5 of both trial arms during the buffet
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
mm
  fasted hunger | 65 (26) | 66 (17)
  fasted fullness | 8 (8) | 21 (17)
  fasted "how much can you eat" | 69 (19) | 65 (20)
  fasted thirst | 93 (10) | 60 (19)
  fasted sweet desire | 42 (29) | 39 (24)
  fasted salt desire | 21 (25) | 42 (27)
  fasted savoury desire | 54 (29) | 67 (22)
  fasted fatty desire | 32 (26) | 45 (21)
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Visual analogue scale for thirst; Test type: Other; p = 0.646, ANOVA; repeated measures
Statistical Analysis 2: Comparison: Hypohydrated vs Rehydrated; visual analogue scale for desire for savoury; Test type: Other; p = 0.403, ANOVA; repeated measures
Statistical Analysis 3: Comparison: Hypohydrated vs Rehydrated; visual analogue scale for desire for salt; Test type: Other; p = 0.022, ANOVA; repeated measures
Statistical Analysis 4: Comparison: Hypohydrated vs Rehydrated; visual analogue scale for hunger; Test type: Other; p = 0.849, ANOVA; repeated measures
Statistical Analysis 5: Comparison: Hypohydrated vs Rehydrated; visual analogue scale for fullness; Test type: Other; p = 0.062, ANOVA; repeated measures
Statistical Analysis 6: Comparison: Hypohydrated vs Rehydrated; visual analogue scale for how much participants felt they could eat; Test type: Other; p = 0.549, ANOVA; repeated measures
Statistical Analysis 7: Comparison: Hypohydrated vs Rehydrated; visual analogue scale for sweet desire; Test type: Other; p = 0.402, ANOVA; repeated measures
Statistical Analysis 8: Comparison: Hypohydrated vs Rehydrated; visual analogue scale for fatty food desire; Test type: Other; p = 0.138, ANOVA; repeated measures

8. Secondary Outcome: Muscle Volume
Description: Comparing muscle size in the dehydrated and rehydrated state.Taken from the pQCT scans
Time Frame: pQCT scans on day 4 of the trial before the dehydration protocol in the heat tent, and on day 5 before the OGTT
Measure: Mean (Standard Deviation); unit: percent change from basline
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
percent change from basline | -2.9 (2.7) | 0.0 (2.1)
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.055, ANOVA — Above is trial*time effect. trial p = 0.135; time p = 0.011; repeated measures

9. Secondary Outcome: Body Water Content
Description: Taken from bioelectrical impedance weighing scales
Time Frame: Daily (i.e. 5 consecutive days for each trial arm)
Measure: Mean (95% Confidence Interval); unit: kg change from baseline
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
kg change from baseline | -0.4 [-0.8 to 0.0] | 0.1 [-0.3 to 0.6]
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p = 0.226, t-test, 2 sided; paired sample

10. Other Pre Specified Outcome: Serum Osmolality
Description: Change from baseline
Time Frame: Measured from the blood samples on day 4 and day 5 on both trial arms
Measure: Mean (Standard Deviation); unit: mosmol/kg
Arm/Group | Hypohydrated | Rehydrated
Number analyzed (Participants) | 16 | 16
mosmol/kg | 9 (6) | 1 (4)
Statistical Analysis 1: Comparison: Hypohydrated vs Rehydrated; Test type: Other; p < 0.001, t-test, 2 sided; paired samples

11. Other Pre Specified Outcome: Plasma Volume
Description: Error in plasma volume measurement during the study invalidated the data
Time Frame: Measured from the blood samples on day 4 and day 5 on both trial arms
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Other Metabolites
Description: Creatinine, cholesterol, triglycerides (if funds allow). No funds, not measured
Time Frame: Collected from the blood samples throughout day 5 of both trial arms
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Muscle Biopsy Measures
Description: These are pilot data for future studies. Muscle glycogen content will be looked at
Time Frame: Using the muscle biopsy samples from participants who opted-in, pre- and post-OGTT on day 5 of each trial
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Psychological Appetite Tests
Description: These are pilot data for future hypotheses looking at subconscious food cues.
Time Frame: Within the 30 minutes before the ad libitum pasta meal
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Hypohydrated | Rehydrated
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes